CLINICAL TRIAL: NCT05606276
Title: Effects of Multi-joint Eccentric Potentiation Maximal Contractions on Muscle Function
Brief Title: Effects of Eccentric Potentiation Activation on Muscle Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Student researcher graduated and study will not be done.
Sponsor: Brennan Thompson (Other)
Responsible Party: Sponsor-Investigator, Brennan Thompson, Associate Professor, Utah State University
Organization: Utah State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 12042c
Record Dates: First submitted 2022-10-24; First posted 2022-11-04 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Post Activation Potentiation

STUDY DESIGN:
Intervention Model Description: Following a familiarization session, subjects will be assigned to an order for performing both an eccentric and a cycle (sham) session (i.e., crossover design, the order being randomized). These will be performed 3-7 days apart.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling exercise (Active Comparator): Cycling on a cycle ergometer instead of doing the experimental eccentric exercise.
  Interventions: Other: Cycle ergometer
- Eccentric exercise (Experimental): Perform 2 sets of maximal eccentric contractions as the single session exercise intervention.
  Interventions: Other: Eccentric Exercise

INTERVENTIONS:
Other: Eccentric Exercise — Individuals will do a randomized crossover intervention involving maximal eccentric contractions (2 sets of 6 per leg; experimental condition)
  Arms: Eccentric exercise
Other: Cycle ergometer — Individuals will do a randomized crossover intervention involving cycling (active control) exercise
  Arms: Cycling exercise

SUMMARY:
The purpose of this study is to examine the potentiation effects of 2 sets of multi-joint eccentric overload maximal contractions on muscle function.

ELIGIBILITY:
Exclusion Criteria:

* lower body surgery or injury in the last 12 months
* have any neuromuscular disease
* height >76 inches tall
* height <54 inches tall
* eccentric strength greater than 725 pounds
* pregnant or plan to be pregnant in the duration of the protocol
* don't do resistance exercise at least once per week
* perform intense cardio or strength training >4 days per week
* Present with any other significant comorbid conditions that would impair the ability to participate in the exercise-based testing

Inclusion criteria:

* 18 - 30 years old
* strength train lower body 1-3 times per week

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Vertical Jump | Baseline (pretest)
  3 countermovement vertical jumps, with 30 seconds of rest between attempts
Vertical Jump | Immediately post intervention
  3 countermovement vertical jumps, with 30 seconds of rest between attempts
Vertical Jump | 12 minutes post intervention
  3 countermovement vertical jumps, with 30 seconds of rest between attempts
Vertical Jump | 20 minutes post intervention
  3 countermovement vertical jumps, with 30 seconds of rest between attempts
Isokinetic eccentric maximal strength | Baseline (pretest)
  Maximal eccentric strength on the Eccentron machine. 2 repetitions per time point
Isokinetic eccentric maximal strength | Immediately post intervention
  Maximal eccentric strength on the Eccentron machine. 2 repetitions per time point
Isokinetic eccentric maximal strength | 12 minutes post intervention
  Maximal eccentric strength on the Eccentron machine. 2 repetitions per time point
Isokinetic eccentric maximal strength | 20 minutes post intervention
  Maximal eccentric strength on the Eccentron machine. 2 repetitions per time point

CONTACTS AND LOCATIONS:
Overall Officials: Brennan J Thompson, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided